CLINICAL TRIAL: NCT06526208
Title: Phase 2 Randomized Placebo-controlled, Double-blind, Parallel Study to Assess the Safety and Efficacy of an Oral Marijuana-Based Investigational Medical Product to Treat Anxiety in Adults With Autism Spectrum Disorder (ASD)
Brief Title: Investigating a Marijuana-based Compound as a Treatment for Anxiety in Autistic Adults
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Southwest Autism Research & Resource Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 168788; RFGA2022-009-001 (Other Grant/Funding Number: Arizona Department of Health Services: ABRC)
Record Dates: First submitted 2024-07-23; First posted 2024-07-29 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Autism Spectrum Disorder; Anxiety
Keywords: Autism; Anxiety; marijuana; cannabis; CBD; THC
MeSH Terms: conditions — Autism Spectrum Disorder; Anxiety Disorders; Autistic Disorder; Marijuana Abuse | interventions — Oils

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MB-IMP Group (Active Comparator): Participants in this group will receive the MB-IMP, an oil-based solution that will contain CBD and THC (23:1 ratio, respectively) and be taken orally. Participants or study partners will dispense the daily dose with an eye dropper according to instructions from the Principal Investigator or delegated study coordinator. Dosing will start at 0.25 ml per day (50 mg of CBD and 2.18 mg of THC). The dose will gradually increase to 1.0 ml per day (200 mg of CBD, and 8.7 mg of TCH) by week 4. Weeks 5 through 8 will be at the maximum dose, 2 ml per day (400 mg of CBD and 17.4 mg of THC). With the exception of week 1 at the lowest dose (0.25 ml), participants will dose in the morning and evening to reach the maximum dose for that time period.
  Interventions: Drug: MB-IMP
- Placebo Group (Placebo Comparator): Participants will follow the same dosing instructions for the MB-IMP group, but will take only MCT oil.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: MB-IMP — MB-IMP is a marijuana-based investigational medical product. It contains a 23:1 ratio of CBD to THC, is an oil-based tincture that is taken orally.
  Other Names: MCT oil
  Arms: MB-IMP Group
Other: Placebo — Does not contain CBD or THC
  Other Names: Medium Chain Triglyceride (MCT) oil
  Arms: Placebo Group

SUMMARY:
The goal of this clinical trial is to learn if drug ABC works to treat severe asthma in adults. It will also learn about the safety of drug ABC. The main questions it aims to answer are:

Will a marijuana-based drug help anxiety in autistic adults?

Anxiety can make socializing and working more difficult for people. Researchers will compare a marijuana based drug (that is mostly CBD with a small amount of THC) to a placebo (a look-alike substance that contains no drug) to see if the drug makes symptoms of anxiety better.

Participants will take the drug (or a placebo) every day for 8 weeks and keep a diary to record the time they took the drug, and their feelings each day. The drug is taken orally in drops once or twice a day. The study staff will speak to the participants weekly either over the phone or in the clinic. Clinic visits once every 2 weeks for checkups and tests. The researchers will make sure participants are healthy and see if there are any changes in anxiety.

DETAILED DESCRIPTION:
The marijuana-based investigation medical product (MB-IMP) in this study is 23 parts CBD and 1 part THC. The placebo is medium chain triglyceride oil. MB-IMP or placebo will be taken orally. DSM-5 diagnosis of autism spectrum disorder will be confirmed with Autism Diagnostic Observation Schedule, version 2, and review of medical records. History of psychosis, suicidality, cardiac or hepatocellular issues may be exclusionary. The participant must have a study partner who will complete observational assessments regarding the participant's behavior.

The screening period is 3 weeks to allow for lab results and medical records to be obtained. The active phase of the study (on drug or placebo) is 8 weeks, and their will be one follow-up visit after 14 days off drug.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female age 18 to 45 years old with an autism diagnosis.
2. Participant is ≥ 100 lbs.
3. Participant or a legally authorized representative provides informed consent/assent for participation in the trial.
4. Participant/caregiver is willing and able to comply with all study procedures.
5. Participant meets ADOS-2 criteria for Autism or Autism Spectrum
6. Participant meets DSM-5 criteria for ASD.
7. Participant has a minimum CGI-S (Anxiety) score ≥ 5 based on anxiety related social functional impairment.
8. Participant has a FSIQ ≥ 65 at screening measured with the WASI- II, or within 1 year of screening with a comparable assessment.
9. Participant must have a negative pregnancy test (urine and serum) at Screening, and a negative urine test at Baseline, Active Phase Visits, and EoS visits, see Table 1. Schedule of Activities.
10. Sexually active participants agree to use two methods of effective birth control, as described in Appendix B: Contraceptive and Barrier Guidance during the study intervention period and for at least 14 days after the Study Termination visit.
11. Participant must be stable on any pre-study medications and/or psychotherapy for 6-weeks prior to study enrollment, agree to inform prescribing clinician(s) about participation in the study, and agree to maintain medication or psychotherapy treatment regimen during the study.
12. Participant must be able to ingest MB-IMP (or placebo) and be willing to commit to medication dosing and completing the dosing diary.
13. Participant/caregiver agrees to keep all study medication provided by site staff securely stored at home and not to share/distribute study medication to any other individual.
14. Participant agrees not to participate in any other interventional clinical trials during the study period.
15. Participant agrees to inform the investigators within 48- hours of any side-effects, medical conditions, and procedures.
16. Participant agrees to abstain from alcohol use during the study.

Exclusion Criteria:

1. Participant weighs < 100 lbs.
2. Participant is sexually active and does not practice two effective forms of birth control.
3. Participant is pregnant, lactating, or planning pregnancy during the study period or within 12 weeks thereafter.
4. Participant has a current or historical psychotic features/disorder assessed via the Mini-International Neuropsychiatric Interview (MINI).
5. Participant has a current or historical DSM-5 diagnosis of dissociative identity disorder, positive family history (first-degree relative) of psychotic disorder or bipolar disorder type 1.
6. At high risk of suicide or suicide attempts.

   1. Individuals presenting current serious suicide risk, as determined through psychiatric interview, responses to the Columbia Suicide Severity Rating Scale (C-SSRS), and/or clinical judgment of the investigator.
   2. History of suicide attempts within 12 months prior to study enrollment.
7. Participant has a current substance use disorder within the 12 months prior to enrollment as determined by the MINI Kid56.
8. Participant's urine drug screen is positive for opiates, methamphetamine, cocaine, THC, and amphetamines (unless prescribed). Participants with positive THC urine analysis tests are excluded from the study but will be allowed to rescreen (maximum twice) after a 1-month cessation of cannabis use.
9. Participant has a history of arrhythmia, other than occasional premature atrial contractions (PACs) and premature ventricular contractions (PVCs) without ischemic heart disease, within 12 months of screening.
10. Participant with a history of atrial fibrillation, atrial tachycardia, atrial flutter or paroxysmal supraventricular tachycardia, or any other arrhythmia associated with a bypass tract, may be enrolled only if they have been successfully treated with ablation and have not had a recurrent arrhythmia for at least one year off all antiarrhythmic drugs or are under adequate and stable pharmacologic treatment for atrial fibrillation for at least a year, as confirmed by a cardiologist.
11. Participant has a current diagnosis or evidence of significant or uncontrolled hematological, endocrine, cerebrovascular, cardiovascular, coronary, pulmonary, gastrointestinal, renal, immunocompromising, or neurological disease according to PI's discretion.
12. Evidence of existing hepatocellular injury defined as alanine transaminase (ALT) and aspertate aminotranferase (AST) elevations of greater than 3 times upper limit normal (ULN) and bilirubin elevation of greater than 2 times ULN.
13. The PI or medical monitor deems the participant inappropriate for the study for any reason.
14. Any known allergies/sensitivities to cannabis (in the opinion of the investigator).
15. Not able to attend required face-to-face visits or those who plan to move out of the area within the treatment period.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 108 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in baseline on reported anxiety related symptoms | 8 weeks
  The Clinical Global Impression Scale for Severity will be used to measure the change in anxiety related symptoms. We hypothesize a two point reduction in severity and

SECONDARY OUTCOMES:
Change in socialization | 8 weeks
  We will measure the Change in behaviors related to socialization with the Social Responsiveness Scale
Change in repetitive behaviors from baseline to the end of study | 8 weeks.
  We will measure the amount of repetitive behaviors with the Repetitive Behavior Scale- Revised
We will measure the change in a variety of aberrant behaviors from baseline to end of study | 8 weeks
  Study partners will complete the Aberrant Behavior Checklist at every clinic visit.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher J Smith, Ph.D., Principal Investigator — SARRC
Locations (1):
- Southwest Autism Research and Resource Center, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No